CLINICAL TRIAL: NCT03334409
Title: Randomized, Phase II Trial of Intravenous Ascorbic Acid (Vitamin C) as an Adjunct to Pazopanib in the First-Line or Post-Immunotherapy Setting for Metastatic or Unresectable Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: Pazopanib Hydrochloride With or Without Ascorbic Acid in Treating Patients With Kidney Cancer That Is Metastatic or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to loss of funding from the private foundation source
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GU-1703; NCI-2017-01998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GU-1703 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v7; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — Ascorbic Acid; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (pazopanib hydrochloride, ascorbic acid) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28 and ascorbic acid IV three times per week. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ascorbic Acid; Drug: Pazopanib Hydrochloride
- Arm B (pazopanib hydrochloride) (Active Comparator): Patients receive pazopanib hydrochloride PO QD on days 1-28. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Drug: Ascorbic Acid — Given IV
  Other Names: 2-(1,2-dihydroxyethyl)-4,5-dihydroxy-furan-3-one; Asorbicap; C Vitamin; C-Long; Ce-Vi-Sol; Cecon; Cenolate; Cetane; Cevalin; L-Ascorbic Acid; VIT C; Vitamin C; Vitamin-C
  Arms: Arm A (pazopanib hydrochloride, ascorbic acid)
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient

SUMMARY:
This randomized phase II trial studies how well pazopanib hydrochloride with or without ascorbic acid work in treating patients with kidney cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Ascorbic acid may help pazopanib hydrochloride stop tumor growth and improve treatment survival. Giving pazopanib hydrochloride and ascorbic acid may work better in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate and compare treatment failure-free rate at 40 weeks from randomization of patients with unresectable/metastatic clear cell renal cell carcinoma (ccRCC) receiving one of the following regimens: Arm A: pazopanib hydrochloride (pazopanib) 800 mg daily plus intravenous (IV) ascorbic acid 1g/kg 3 times/week and Arm B: pazopanib 800 mg daily.

SECONDARY OBJECTIVES:

I. To estimate and compare the overall survival (OS) in patients receiving pazopanib with or without IV ascorbic acid.

II. To estimate and compare the progression-free survival (PFS) in patients receiving pazopanib with or without IV ascorbic acid.

III. To estimate and compare the overall response rate (ORR) in patients receiving pazopanib with or without IV ascorbic acid.

IV. To estimate and compare the duration on pazopanib treatment in patients receiving pazopanib with or without IV ascorbic acid.

V. To assess the adverse events (AE) profile and safety of each treatment arm using the Common Terminology Criteria for Adverse Events (CTCAE).

CORRELATIVE RESEARCH:

I. Correlation between 5 mC, 5 hmC and H3K27me3 expression (as determined by immunohistochemistry [IHC]), as well as MeDIP/hMeDIP sequencing (seq), and response to combination of IV ascorbic acid and pazopanib.

II. Correlation between iron content in tumor microenvironment (as determined by Prussian blue staining) and response to combination of IV ascorbic acid and pazopanib combination.

III. Correlation between HIF-1alpha and HIF-2alpha expression (as determined by immunohistochemistry [IHC]) and response to combination of IV ascorbic acid and pazopanib combination.

IV. Correlation between GLUT1 expression (as determined by IHC) and response to combination of IV ascorbic acid and pazopanib.

V. Correlation between PDL1 expression (as determined by IHC) and response to combination of IV ascorbic acid and pazopanib.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28 and ascorbic acid IV three times per week. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive pazopanib hydrochloride PO QD on days 1-28. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of clear cell renal cancer
* Documented metastatic or unresectable disease and at least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) criteria; NOTE: Nephrectomy or ablation of the primary tumor is allowed prior to enrollment
* No prior systemic therapy for clear cell renal cancer or have progressed after immunotherapy such as ipilimumab plus nivolumab in the first line; other immunotherapies (e.g. interleukin-2) or additional lines of immunotherapy may be allowed after discussion with the principal investigator
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 21 days prior to registration)
* Platelet (PLT) >= 100,000/mm^3 (obtained =< 21 days prior to registration)
* Hemoglobin (Hgb) >= 9.0 g/dL (obtained =< 21 days prior to registration); NOTE: Subjects may not have had a transfusion =< 7 days of registration
* Total Bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 21 days prior to registration)

  * NOTE: For bilirubin elevation 1 to 1.5 x ULN, alanine aminotransferase (ALT) above 1.5 x ULN (upper limit of normal) is not permitted
  * NOTE: For bilirubin elevation 1 to 1.5 x ULN, aspartate aminotransferase (AST) above 1.5 x ULN (upper limit of normal) is not permitted
* Alanine amino transferase (ALT) < 2.5 X ULN, with normal bilirubin (obtained =< 21 days prior to registration); NOTE: Concomitant elevations in bilirubin and ALT above 1.5 x ULN (upper limit of normal) is not permitted
* Aspartate aminotransferase (AST) < 2.5 X ULN, with normal bilirubin (obtained =< 21 days prior to registration); NOTE: Concomitant elevations in bilirubin and AST above 1.5 x ULN (upper limit of normal) is not permitted
* Creatinine =< 1.5 mg/dl OR creatinine > 1.5 mg/dl, estimated creatinine clearance must be >= 55 mL/minute by Cockcroft Gault formula (obtained =< 21 days prior to registration)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (obtained =< 21 days prior to registration); NOTE: This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose
* Individuals of non-childbearing potential, or individual of childbearing potential with negative serum pregnancy test =< 7 days prior to randomization and willing to practice total abstinence or use a highly effective method of contraception, as outlined below:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female individual who has had the following:

    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal
    * NOTE: Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40 pg/mL (< 140 pmol/L); subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
  * Childbearing potential, including any individual who has had a negative serum pregnancy test, =< 7 days prior to randomization
  * Agrees to use adequate contraception; acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
    * Oral contraceptive, either combined or progestogen alone
    * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
    * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
    * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Provide informed written consent
* Willing to provide archive tissue samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Individuals/or persons who are nursing
  * Individual/or persons who are pregnant
  * Individuals/or persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Prior history of receiving pazopanib or any other tyrosine kinase inhibitor treatments for malignancy
* Uncontrolled intercurrent illness including, but not limited to:

  * Chronic ongoing or active infection
  * Symptomatic anemia
  * Uncontrolled hypertension (defined as systolic blood pressure [SBP] of >= 160 mmHg or diastolic blood pressure [DBP] of >= 100 mmHg)
  * Symptomatic congestive heart failure as defined by the New York Heart Association (NYHA) (does not exclude class III congestive heart failure [CHF])
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Evidence of active bleeding or bleeding diathesis
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other serious uncontrolled medical disorders in the opinion of the investigator
* History of a major thromboembolic event =< 6 months prior to randomization, including cerebrovascular accident, transient ischemic attack (TIA), myocardial infarction, symptomatic pulmonary embolism (PE) or untreated deep venous thrombosis (DVT), or coronary artery bypass graft surgery; NOTE: Subjects with recent DVT or asymptomatic PE who have been treated with therapeutic anticoagulating agents for at least 6 weeks are eligible
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to randomization; EXCEPTIONS: Nonmelanoma skin cancer or carcinoma-in-situ of the cervix, or cancers with low metastatic potential (e.g. Gleason score 6 prostate cancer) treated with curative therapy; NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for =< 6 months prior to randomization; Note: Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn?s disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 28 days prior to randomization
  * Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

    * Malabsorption syndrome
    * Any prior major resection of the stomach or small bowel
* Corrected QT interval (QTc) > 480 msecs using Bazett?s formula
* Receiving any medications or substances with risk of Torsades de Pointes; Note: medications or substances on the list ?Drugs with Risk of Torsades de Pointes? are prohibited; medications or substances on the list ?Drugs with Possible or Conditional Risk of Torsades de Pointes? may be used while on study with extreme caution and careful monitoring
* Treatment with any of the following anti-cancer therapies =< 14 days prior to registration:

  * Radiation therapy
  * Surgery or tumor embolization
  * Chemotherapy, immunotherapy
  * Biologic therapy
  * Investigational therapy
  * Hormonal therapy
* Prior autologous or allogeneic organ or tissue transplantation
* Elective or planned major surgery to be performed during the course of the trial
* Receiving any medications or substances that are strong or moderate inhibitors of CYP3A4; use of strong or moderate inhibitors are prohibited =< 7 days prior to randomization
* Receiving any medications or substances that are inducers of CYP3A4; use of inducers are prohibited =< 7 days prior to randomization
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency (i.e. below normal limits)
* End-stage renal disease (estimated glomerular filtration rate [GFR] < 55 ml/min/body surface area [BSA]), unless the estimated creatinine clearance by Cockcroft Gault is >= 55 ml/min prior to randomization
* History of calcium oxalate stones
* History of iron overload
* Unable to swallow oral medications
* History of myocardial infarction =< 6 months, current symptomatic CHF or left ventricular ejection fraction (LVEF) < 40% or > grade 2 diastolic dysfunction, with no symptoms or signs of heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance C Pagliaro, Principal Investigator — Academic and Community Cancer Research United
Locations (5):
- United States (5):
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Sanford Medical Center Fargo, Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Started | 2 | 3
Completed | 1 | 3
Not Completed | 1 | 0
Not completed — Did not meet inclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride) | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 55 [55 to 55] | 56.7 [47.0 to 68.0] | 56.3 [47 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
MSKCC Risk Factor [Count of Participants; unit: Participants] — For each of the following criteria answered as 'Yes', 1 point is assigned: ECOG Performance Status >=2; Corrected Calcium >10 mg/dl (≥ 2.5 mmol/L); Hemoglobin less than the lower limit of normal - where the normal range for hemoglobin are between 13.5 and 17.5 g/dl for men and between 12.0 and 15.5 g/dl for women; Time from diagnosis to systemic treatment < 1year (previously untreated patients only); Lactate dehydrogenase > 1.5x upper limit of normal - where the upper normal is 140U/L (previously untreated patients only). Total of 0 = Favorable risk, 1-2 = Intermediate risk, 3 >= Poor risk
  Participants
    Poor risk | 1 | 1 | 2
    Intermediate risk | 0 | 1 | 1
    Favorable risk | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure-free Rate
Description: Treatment failure is defined as any of the following: radiographic disease progression, off-protocol treatment due to adverse event, initiation of alternative therapy (except metastasectomy post clinical benefit (complete response [CR], partial response [PR], or stable disease [SD] per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 to treatment), and death due to any cause.
Time Frame: At 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Number analyzed (Participants) | 1 | 3
Participants | 0 | 2
Statistical Analysis 1: Comparison: Arm A (Pazopanib Hydrochloride, Ascorbic Acid) vs Arm B (Pazopanib Hydrochloride); Test type: Superiority; p = 1.0, Fisher Exact

2. Secondary Outcome: Overall Survival
Description: Will be estimated using the method of Kaplan-Meier and be compared using log rank tests.
Time Frame: 26 months
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Number analyzed (Participants) | 1 | 3
Months | 7.8 [NA to NA] — Too few patients to calculate. | NA [NA to NA] — No events occurred, the lower limit, median, and upper limit were not reached.
Statistical Analysis 1: Comparison: Arm A (Pazopanib Hydrochloride, Ascorbic Acid) vs Arm B (Pazopanib Hydrochloride); Test type: Superiority; p = 0.08, Log Rank

3. Secondary Outcome: Progression Free Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: 16 Months
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Number analyzed (Participants) | 1 | 3
Months | 5.7 [5.7 to 5.7] | 11.8 [7.3 to 15.9]
Statistical Analysis 1: Comparison: Arm A (Pazopanib Hydrochloride, Ascorbic Acid) vs Arm B (Pazopanib Hydrochloride); Test type: Superiority; p = 0.08, Log Rank

4. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan, PET/CT, or MRI: Complete Response (CR), Disappearance of all target lesions and all target lymph nodes must have reduction in short axis to <1.0 cm; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation; Overall Response (OR) = CR + PR. Will be compared using a Chi-Square test.
Time Frame: 16 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Number analyzed (Participants) | 1 | 3
Participants | 0 | 1
Statistical Analysis 1: Comparison: Arm A (Pazopanib Hydrochloride, Ascorbic Acid) vs Arm B (Pazopanib Hydrochloride); Test type: Superiority; p = 1, Fisher Exact

5. Secondary Outcome: Duration of Time on Pazopanib Hydrochloride
Description: Will be described as the median time on treatment by arm.
Time Frame: 10 months
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Number analyzed (Participants) | 1 | 3
Months | 5.9 [5.9 to 5.9] | 9.2 [7.3 to 9.2]
Statistical Analysis 1: Comparison: Arm A (Pazopanib Hydrochloride, Ascorbic Acid) vs Arm B (Pazopanib Hydrochloride); Test type: Superiority; p = 0.18, Kruskal-Wallis

6. Secondary Outcome: Frequency of Adverse Events
Description: Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Adverse events and toxicities will be evaluated using all patients who have received any study treatment as well as summarizing those who have been included in the efficacy analyses. The overall adverse event frequencies for grade 3 or higher adverse events, will be compared using Chi-Square tests between the 2 treatment arms.
Time Frame: 10 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
Number analyzed (Participants) | 1 | 3
Participants | 1 | 2
Statistical Analysis 1: Comparison: Arm A (Pazopanib Hydrochloride, Ascorbic Acid) vs Arm B (Pazopanib Hydrochloride); Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed up to 10 months. All-Cause Mortality assessed up to 26 months
Arm/Group | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) | Arm B (Pazopanib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) (N=1) | Arm B (Pazopanib Hydrochloride) (N=3)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Pazopanib Hydrochloride, Ascorbic Acid) (N=1) | Arm B (Pazopanib Hydrochloride) (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (19)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (4) | 3 (15)
Fatigue (General disorders) | 1 (6) | 3 (26)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (3)
Pain (General disorders) | 0 (0) | 1 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 2 (15)
GGT increased (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 0 (0) | 1 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (8)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (4) | 3 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03334409/Prot_SAP_000.pdf